CLINICAL TRIAL: NCT01116362
Title: Study of Surgical Methods for Repair of Clean Transections in Peripheral Nerve Injuries
Brief Title: Comparing Primary With Secondary Repair of Based on Electrodiagnostic Assessment and Clinical Examination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy/Associate Professor of Medical Education, Isfahan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-1213-2
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2008-03

CONDITIONS: Peripheral Nerve Injury
Keywords: ulna; median; repair; primary
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- secondary repair (Other): secondary closure beyond the first week.the nerve was conducted to repair as end to end (epi-epineurium, epi-epineurium) anastomosis. This was performed following the repair of present tendons and muscle injuries.
  Interventions: Procedure: secondary repair
- primary repair (Other): during first days,the nerve was conducted to repair as end to end (epi-epineurium, epi-epineurium) anastomosis. This was performed following the repair of present tendons and muscle injuries.
  Interventions: Procedure: primary repair

INTERVENTIONS:
Procedure: primary repair — during the first days,the nerve was conducted to repair as end to end (epi-epineurium, epi-epineurium) anastomosis. This was performed following the repair of present tendons and muscle injuries.
  Other Names: NCV,EMG
  Arms: primary repair
Procedure: secondary repair — after one week,the nerve was conducted to repair as end to end (epi-epineurium, epi-epineurium) anastomosis. This was performed following the repair of present tendons and muscle injuries.
  Other Names: NCV,EMG
  Arms: secondary repair

SUMMARY:
The purpose of this study is to determine which surgical approach is better for clean transection injury in peripheral nerves in outcomes.

DETAILED DESCRIPTION:
Treatment of injuries to major nerve trunks in the hand and upper extremity remains a major and challenging reconstructive problem. Our goal was to compare primary versus secondary repair of median and\or ulnar nerve by electrodiagnostic assessment and clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed clean transection injury between shoulder and wrist

Exclusion Criteria:

* crush injuries

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
motor function | at 18 months post-operatively
  identification of motor level were done based on British Medical Research Council guided.The abductor pollicis brevis (APB) was used for the median nerve and the abductor digiti minimi (ADM) for the ulnar nerve. as follows: 0, M0, M1 and M2; 1, M3; 2, M4.

SECONDARY OUTCOMES:
sensory recovery | at 18 months post-operatively
  identification of motor and sensory level were done based on British Medical Research Council guided.The abductor pollicis brevis (APB) was used for the median nerve and the abductor digiti minimi (ADM) for the ulnar nerve. The results scored as follows: 0, S0, S1 and S2; 1, S3; 2, S4 and S5.
nerve conduction velocity | at 18 months post-operatively
  For electrodiagnostic assessment, nerve conduction velocity (NCV) was tested as motor and sensory. The results categorized according to the Yale sensory scale and the severity of sensation and function of the nerves was scored as follows: 0, no sensation; 1, decreased or abnormal sensation; 2, normal sensation.
electromyography | at 18 months post-operatively
  For an EMG, a needle electrode was inserted through the skin into the muscle which injured nerve supplied. The presence, size and shape of the waveform registered and the ability of the muscle to respond when the nerves were stimulated. Also these results scored as follows: 0, no activity; 1, few or single movement; 2, partial activity; 3, full activity.

CONTACTS AND LOCATIONS:
Overall Officials: hamidreza shemshaki, MD, Study Chair — MD,research comittee
Locations (1):
- Al-zahra university hospital, Isfahan, Iran